CLINICAL TRIAL: NCT02467114
Title: Interactions Between Attentional Networks and Their Influence on Perception: a Project in Healthy Subjects and Hemispatial Neglect Patients
Brief Title: Interactions Between Attentional Networks and Their Influence on Perception
Acronym: AtNet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 036/15
Record Dates: First submitted 2015-05-27; First posted 2015-06-09 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Stimulation with TMS, a sham coil & no intervention
  Interventions: Device: Transcranial magnetic stimulation (TMS); Device: Sham coil stimulation; Other: Control without stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — This method will be applied to measure cortical excitability and as an interference approach; real TMS stimulation will be compared with sham stimulation and no stimulation
Device: Sham coil stimulation — Stimulation with a sham coil as a comparison
Other: Control without stimulation

SUMMARY:
Attention can be defined as the preparedness to rapidly and accurately respond to stimuli coming from the investigators environment and to effectively select between relevant and irrelevant information. According to a current model, visual attentional control is based on two separate groups of brain regions, so called brain networks. These networks control different attentional aspects (e.g., spatial/non-spatial attention) and they interact with each other. A disruption of these interactions can lead to attentional disorders such as hemispatial neglect. Patients with hemispatial neglect have difficulties directing their attention to the left visual field and they act as though the latter does not exist.

To date, the interactions between the two attentional networks are poorly understood. The aim of this study consists in further clarifying different aspects of these interactions and their influence on visual perception in healthy participants and in patients with hemispatial neglect. Transcranial magnetic stimulation (TMS) will be the principal method applied in this study. TMS is a painless and non-invasive method, with which the activity of brain areas can be influenced temporarily. This allows us to draw conclusions regarding the functions and interactions of these brain areas.

This study is designed to have a significant impact on the basic understanding of attentional control in the human brain and it can benefit the comprehension and treatment of attentional disorders, such as hemispatial neglect.

DETAILED DESCRIPTION:
Background

Attention can be defined as the preparedness to rapidly and accurately respond to stimuli coming from the investigators environment and to effectively select between relevant and irrelevant information. Attention is a complex cognitive function based on multiple components. A recent model postulates that attentional control in the brain is based on two discrete neural networks. The ventral (temporo-parietal - ventral frontal) network controls non-spatial aspects of attention, such as alertness and vigilance, and stimulus detection and reorientation in both hemifields. This network is lateralized towards the right hemisphere and plays a role as a 'circuit-breaker'. The dorsal (superior parietal - dorsal frontal) network controls spatial attentional shifts, is largely top-down driven, and substantially overlaps with eye movement control. This network is not functionally lateralized, each hemisphere containing dynamic topographical maps of the contralateral space. Moreover, the dorsal networks of the two hemispheres compete to direct attention to the contralateral hemispace, thereby exerting reciprocal inhibition.

Hemispatial neglect - the failure to detect, orient, or respond to stimuli located in the contralesional side of space - has been interpreted in terms of pathological changes in the interaction between the two attentional networks. Neglect is very common after cerebral lesions of the right hemisphere, usually affecting the ventral attentional network. The structurally intact right dorsal network would thus receive a weakened input from the right ventral network. The ensuing imbalance in the inhibition between the dorsal networks of the two hemispheres would then result in the rightward bias in attentional allocation, typically observed in hemispatial neglect.

However, little is known regarding the interactions between ventral and dorsal attentional networks and their influence on perception, and the greatest part of the evidence has been acquired through correlational approaches. The aim of this study is to further elucidate different aspects of these interactions and to investigate their influence on spatial and non-spatial attentional performance and on visual perception.

Objective

A first objective consists in further elucidating how and through which anatomical structures the ventral and the dorsal attentional networks interact. A second objective concerns how the interplay of dorsal and ventral attentional networks influences visual perception, in particular in cases in which visual stimuli are ambiguous.

Methods

Transcranial magnetic stimulation (TMS) is the principal method applied in this study. TMS is a non-invasive, painless method which is able to influence cortical areas directing attention in an interference approach and to thus establish causal relationships. Furthermore, TMS, in combination with the measurement of motor evoked potentials (MEP), allows for the assessment of the excitability of cortico-cortical circuits.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy participants:
* Age 18-80 years
* Neurologically healthy, i.e., with no documented or present neurological disease or brain injury
* normal or corrected-to-normal visual acuity
* Patients:
* Age 18-80 years
* Showing signs of left hemispatial neglect after a right-hemispheric brain lesion, as assessed by previous neuropsychological testing and clinical judgment
* Normal or corrected-to-normal visual acuity

Exclusion Criteria

* Healthy participants:
* Any instable medical condition, in particular epilepsy (past or present, including seizures or febrile convulsions)
* Any surgical intervention to the brain
* Implanted medical devices (e.g., cochlear implants, infusion pumps, neurostimulators, pacemakers)
* Presence of metal in the region of the head (excluding fixed dental implants such as tooth fillings or fixed dental braces)
* Drug or alcohol abuse
* Intake of any medication that is likely to lower seizure threshold
* For female participants: pregnancy or breast feeding or intention to become pregnant during the course of the experiment. All participants of childbearing potential will be asked to take a pregnancy test.
* Patients:
* Any instable medical condition, in particular epilepsy (past or present, including seizures or febrile convulsions)
* Implanted medical devices (e.g., cochlear implants, infusion pumps, neurostimulators, pacemakers)
* Presence of metal in the region of the head (excluding fixed dental implants such as tooth fillings or fixed dental braces)
* Drug or alcohol abuse
* Intake of any medication that is likely to lower seizure threshold
* For female participants: pregnancy or breast feeding or intention to become pregnant during the course of the experiment. All participants of childbearing potential will be asked to take a pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Cortical excitability, as measured by motor evoked potentials (MEPs) | During or within 1 hour after application
Spatial attentional performance, as measured by cognitive testing | During or within 1 hour after application
Number of perceptual switches | During or within 1 hour after application
Duration of dominance phases of perceptual switches | During or within 1 hour after application
  Measured in seconds

SECONDARY OUTCOMES:
Alertness level, as measured subjectively by a visual analogue scale (VAS) | During or 1 hour after application
Alertness level, as measured objectively by cognitive testing | During or 1 hour after application
Spatial bias of attentional allocation, as measured by standardised paper-pencil neuropsychological tests | During or 1 hour after application
Spatial bias of attentional allocation, as measured by free visual exploration with eye movement measurement | During or 1 hour after application

CONTACTS AND LOCATIONS:
Overall Officials: René M. Müri, Prof. Dr. med., Principal Investigator — Department of Neurology, Inselspital, Bern University Hospital; Thomas Nyffeler, Prof. Dr. med., Principal Investigator — Center for Neurology and Neurorehabilitation, Luzerner Kantonsspital
Locations (1):
- Division of Cognitive and Restorative Neurology, Department of Neurology, Inselspital, Bern University Hospital; Gerontechnology and Rehabilitation Group, ARTORG Center for Biomedical Engineering Research, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Corbetta M, Patel G, Shulman GL. The reorienting system of the human brain: from environment to theory of mind. Neuron. 2008 May 8;58(3):306-24. doi: 10.1016/j.neuron.2008.04.017. PMID 18466742
- [Background] Corbetta M, Shulman GL. Control of goal-directed and stimulus-driven attention in the brain. Nat Rev Neurosci. 2002 Mar;3(3):201-15. doi: 10.1038/nrn755. PMID 11994752
- [Background] Corbetta M, Shulman GL. Spatial neglect and attention networks. Annu Rev Neurosci. 2011;34:569-99. doi: 10.1146/annurev-neuro-061010-113731. PMID 21692662
- [Background] Koch G, Oliveri M, Cheeran B, Ruge D, Lo Gerfo E, Salerno S, Torriero S, Marconi B, Mori F, Driver J, Rothwell JC, Caltagirone C. Hyperexcitability of parietal-motor functional connections in the intact left-hemisphere of patients with neglect. Brain. 2008 Dec;131(Pt 12):3147-55. doi: 10.1093/brain/awn273. Epub 2008 Oct 22. PMID 18948300
- [Background] Sack AT. Using non-invasive brain interference as a tool for mimicking spatial neglect in healthy volunteers. Restor Neurol Neurosci. 2010;28(4):485-97. doi: 10.3233/RNN-2010-0568. PMID 20714073